CLINICAL TRIAL: NCT07374796
Title: Signature Development and Validation Protocol for an Epigenetic Assay in Diagnosing Breast Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: EPOCH Epigenetics, Inc (Unknown)
Responsible Party: Principal Investigator, Peter Olivieri, Chair, Division of Pulmonary & Critical Care; Director, Interventional Pulmonary Program, University of Maryland, Baltimore
Other Study IDs: HP-00117656
Record Dates: First submitted 2026-01-20; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer (Locally Advanced or Metastatic); Healthy Volunteers (HV); Unhealthy Volunteers; Breast Cancer Screening
Keywords: Breast Cancer; Breast Cancer Screening; Healthy Volunteers; Unhealthy Volunteers
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral Blood Mononuclear Cells (PBMC)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Study Population 1: This study population will consist of individuals who have a diagnosis of breast cancer and have not received chemotherapy treatment for their breast cancer. Individuals who have received surgical resection and/or radiation therapy and/or endocrine therapy for their breast cancer will be included.
  Interventions: Other: Epigenetic Assay
- Study Population 2: This study population will consist of individuals who have a diagnosis of breast cancer and have received chemotherapy treatment for their breast cancer. All stages of breast cancer will be included including individuals in remission.
  Interventions: Other: Epigenetic Assay
- Study Population 3: This study population will consist of individuals who are at high risk of developing breast cancer.
  Interventions: Other: Epigenetic Assay

INTERVENTIONS:
Other: Epigenetic Assay — Up to 15 ml of blood will be collected from each patient at various time points throughout their 5 years of participation. DNA extraction, bisulfite conversion and analysis of epigenetic markers through PCR or next-generation sequencing will be performed. An epigenetic signature assay will then be identified.

SUMMARY:
The purpose of this research study is to test a new process for diagnosing breast cancer by examining changes to your DNA that can be detected from a blood test. The information we learn by doing this study could potentially help people in the future.

Participants in this study will have blood samples collected, have their medical records reviewed by study personnel and fill out questionnaires at different time points during the study. Blood sample collection will occur during normal routine clinic visits. Participation in this study will last approximately 5 years.

DETAILED DESCRIPTION:
This clinical testing protocol outlines the validation process for an epigenetic assay targeting host peripheral blood cell and the associated host DNA methylation signatures designed to diagnose breast cancer. The overall protocol process will involve three distinct stages representing three patient cohorts with up to 150 subjects per cohort across 3 populations of patients. Cohort one will act as signature development phase; cohort two will act as signature finalization phase; and cohort three will act as a validation cohort phase. Each cohort with include the following patient populations with up to 50 patients per population:

1. Breast cancer, NO chemotherapy. Includes patients treated with surgical resection and/or radiation therapy and/or endocrine therapy
2. Breast cancer who have received chemotherapy. Includes all stages including remission
3. At risk group (patients at increased risk for breast cancer followed in a high risk breast program)

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* Patient of UMMS
* Willing and able to consent to study procedures listed in the protocol
* Ability to speak and understand English

Exclusion Criteria:

* Younger than 18 years old
* Patient not cared for at UMMS
* Unable to consent to study procedures listed in the protocol
* Unable to speak or understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study participants will be selected from patients being cared for across the University of Maryland Medical System
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2032-03 (Estimated); Study Completion 2032-04 (Estimated)

PRIMARY OUTCOMES:
Identification of tumor-associated host methylation signature | 5 years
  Genome-wide methylation profile of whole blood from lung cancer patients, pre-cancer patients, patients undergoing therapy, and control subjects.
Technology development | 5 years
  The investigators will develop array-based assays using whole-blood samples, focused on disease-specific methylation sites to provide early diagnosis, prognosis, and therapeutic efficacy prediction.
Technology validation | 5 years
  The investigators will validate identified blood-based circulating methylation signatures in patients with undiagnosed pulmonary nodules.

SECONDARY OUTCOMES:
EORTC QLQ-C30 Questionnaire | 5 years
  The European Organization for Research and Treatment of Cancer core quality of life questionnaire, (EORTC QLQ-C30) is a cancer-specific quality of life instrument designed to assess health-related quality of life of cancer patients and is intended to be supplemented by disease-specific questionnaires, such as the lung cancer specific module, the EORTC QLQ-LC13. The EORTC QLQ-C30 incorporates nine multi-item scales including five functional scales (Physical, Role, Cognitive, Emotional and Social Functioning); three symptom scales (Fatigue, Pain and Nausea/Vomiting); and a Global Health Status/QoL scale. Six single item scales are also included (Dyspnea, Insomnia, Appetite Loss, Constipation, Diarrhea and Financial Difficulties). All of the scales and single-item measures range in score from 0 to 100. A higher score represents a higher level of symptom burden.
EORTC QLQ-BR45 Questionnaire | 5 years
  EORTC QLQ-BR45 is a supplementary questionnaire module to be employed in conjunction with the QLQ-C30. The QLQ-BR45 incorporates nine multi-item scales to assess body image, sexual functioning, breast satisfaction, systemic therapy side effects, arm symptoms, breast symptoms, endocrine therapy symptoms, skin mucosis symptoms, endocrine sexual symptoms. In addition, single items assess sexual enjoyment, future perspective and being upset by hair loss. All of the scales and single item measures range in score from 0 to 100. A high score for the functional scales and functional single items represents a high/healthy level of functioning, whereas a high score for the symptom scales and symptom item represents a high level of symptomatology or problems.
SF-36v2 Questionnaire | 5 years
  The short-form of 36 questions (SF-36v2) is a multipurpose, 36-item survey that measures eight domains of health: physical functioning, role limitations due to physical health, bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems, and mental health. It yields scale scores for each of these eight health domains, and two summary measures of physical and mental health. Higher scores indicate better health status.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland Baltimore Washington Medical Center, Glen Burnie, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li Y, Fan Z, Meng Y, Liu S, Zhan H. Blood-based DNA methylation signatures in cancer: A systematic review. Biochim Biophys Acta Mol Basis Dis. 2023 Jan 1;1869(1):166583. doi: 10.1016/j.bbadis.2022.166583. Epub 2022 Oct 18. PMID 36270476